CLINICAL TRIAL: NCT06928220
Title: A Single-Center, Prospective, Randomized Clinical Trial Investigating the Impact of Manual Versus Mechanical Intestinal Suturing on the Incidence and Management of Postoperative Complications in Patients Undergoing Radical Cystectomy With Ileal Conduit.
Brief Title: The Impact of Manual Versus Mechanical Intestinal Suturing on the Incidence of Postoperative Complications Following Cystectomy With Ileal Conduit
Acronym: CIMMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio Puigvert (Other)
Responsible Party: Principal Investigator, Pavel Gavrilov, Consultant surgeon, Fundacio Puigvert
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 181184
Record Dates: First submitted 2021-01-18; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Bladder Cancer; Anastomosis; Complications; Ileus Paralytic
Keywords: bladder Cancer; Cystectomy; hand sewn anastamosis; stapled anastamosis; intestinal complications
MeSH Terms: conditions — Urinary Bladder Neoplasms; Ileus | interventions — Cystectomy; Urinary Diversion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual anastamosis (Active Comparator): Intestinal anastamosis will be performed manually
  Interventions: Procedure: cystectomy with ileal conduit, using manual bowel anastomosis
- Mechanical anastamosis (Active Comparator): Intestinal anastamosis will be performed using stapling device
  Interventions: Procedure: cystectomy with ileal conduit, using mechanical bowel anastomosis

INTERVENTIONS:
Procedure: cystectomy with ileal conduit, using mechanical bowel anastomosis — An ileal conduit will be the new storage area for urine once the bladder is removed.
  GIA Device will be used to perform bowel anastomosis
  Arms: Mechanical anastamosis
Procedure: cystectomy with ileal conduit, using manual bowel anastomosis — An ileal conduit will be the new storage area for urine once the bladder is removed.
  Vycryl suture will be used to perform manual bowel anastomosis
  Arms: Manual anastamosis

SUMMARY:
Impact of Manual Versus Mechanical Intestinal Suturing on the Incidence and Management of Postoperative Complications in Patients Undergoing Radical Cystectomy with Ileal Conduit.

DETAILED DESCRIPTION:
Currently, no specific trial compares hand-sewn intestinal anastomosis with mechanical stapled anastomosis in patients undergoing radical cystectomy with ileal conduit.

At Fundació Puigvert, approximately one hundred radical cystectomies with ileal conduit are performed annually. Due to the lack of evidence regarding the superiority of either intestinal anastomosis technique, the decision to use hand-sewn versus stapled anastomosis depends on the surgeon's expertise, without considering the potential impact of each technique on postoperative complication rates, surgical time, or functional outcomes.

Currently, no well-designed surgical trials demonstrate differences between hand-sewn and mechanical stapled anastomosis in radical cystectomy regarding intraoperative and postoperative complications. For this reason, the investigators will conduct a trial to assess the impact of each anastomosis technique

ELIGIBILITY:
Inclusion Criteria:

* Patient who consents to participate and signs the informed consent.
* Patient candidate for radical open cystectomy and ileal conduit.

Exclusion Criteria:

* Patient who is unable to complete the study questionnaires.
* Patient who has a life expectancy of less than 1 year.
* Candidate patients for other urinary diversions other than ileal conduit as a first option
* Candidate patients for laparoscopic or robotic cystectomy..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Demonstrate the superiority of manual intestinal suturing versus mechanical suturing, defined as a lower incidence of postoperative digestive complications in patients undergoing radical cystectomy with ileal conduit. | 1 year
  Compare the incidence of gastrointestinal complications according to the type of suturing used in the creation of the ileo-ileal anastomosis in patients undergoing radical cystectomy with ileal conduit during the hospital admission period and at one-year follow-up.

SECONDARY OUTCOMES:
To evaluate the predictive factors of postoperative complications. | 1 year
  Identify the predictive factors of postoperative complications during hospital admission and at one-year follow-up, both overall and according to the type of suturing.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundacio Puigvert, Barcelona, Barcelona, Spain